CLINICAL TRIAL: NCT05352412
Title: Piloting a Shared Decision-Making Aid for Reducing Stigma in Drug Use and HIV Harm Reduction in a Rural Setting
Brief Title: Stigma and a Shared Decision Aid
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 202107155
Record Dates: First submitted 2022-04-18; First posted 2022-04-28 (Actual); Results first posted 2025-06-24 (Actual); Last update posted 2025-06-24 (Actual); Status verified 2025-06

CONDITIONS: Opioid Use Disorder
Keywords: Stigma; Decision Aid
MeSH Terms: conditions — Opioid-Related Disorders; Social Stigma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Baseline Counseling As Usual - Patient (No Intervention): Patients randomized to the baseline counseling from their healthcare provider regarding medications for opioid use disorder.
- Shared Decision Making Aid - Patient (Active Comparator): Patients randomized to the decision aid arm will receive all of the above as well as a shared decision making aid. This will be a 10-minute survey that takes into account their priorities and preferences around medications for opioid use disorder.
  Interventions: Behavioral: Shared Decision Making Aid - Patients
- Baseline Counseling As Usual - Provider (No Intervention): Providers of patients randomized to the baseline counseling as usual arm will will be asked to participate in a survey to assess their stigma in regards to taking care of patients with opioid use disorder.
- Shared Decision Making Aid - Provider (Active Comparator): Providers of patients randomized to the decision aid arm will will be asked to participate in a survey to assess their stigma in regards to taking care of patients with opioid use disorder.
  Interventions: Behavioral: Shared Decision Making Aid - Providers

INTERVENTIONS:
Behavioral: Shared Decision Making Aid - Patients — Patients will be randomized to the shared decision making aid intervention.
  Arms: Shared Decision Making Aid - Patient
Behavioral: Shared Decision Making Aid - Providers — Providers of patients randomized o the shared decision making aid intervention.
  Arms: Shared Decision Making Aid - Provider

SUMMARY:
A major barrier for the uptake of evidence-based interventions to address the ongoing opioid epidemic in the US, especially in rural regions, is stigma, which occurs at many levels, including that of the patient and provider. A shared decision making aid is an evidence-based method for increasing engagement and knowledge of both patients and providers, potentially democratizing treatment decisions, especially in stigmatized conditions. The investigators propose to adapt and pilot a decision aid for opioid use disorder (OUD) treatment and harm reduction in two hospitals in rural Missouri to evaluate whether this reduces stigma in both patients and providers.

DETAILED DESCRIPTION:
In the past decade, the US opioid crisis has emerged as a leading cause of death among adults. It has also led to an increase in invasive bacterial and fungal infections; and HIV and hepatitis C virus (HCV) outbreaks in multiple regions. Rural communities have had an especially disproportionate burden from the impact of opioid use disorder (OUD). Treatment of OUD with pharmacotherapy is one of the most effective strategies for reducing OUD-related mortality and morbidity. But while there has been increasing will for expanding pharmacotherapy, stigma - from community, providers and patients-remains a significant barrier to uptake pharmacotherapy and harm reduction. The approach to substance use has historically favored abstinence strategies that are often without evidence, influenced by punitive, stigmatizing framework. This stigma may be even more prevalent in rural communities. To date there have been very few effective interventions to address inter- and intrapersonal stigma, and none with sustained effectiveness. The investigators propose adapting and piloting a shared decision-making aid for patients presenting to the emergency department or are being admitted at two hospitals in rural Missouri, where there is a high prevalence of OUD and its complications. The decision-aid is an evidence-based intervention show to increase knowledge, engagement and decision-making concordant with patient values in a variety of medical conditions. It is feasible that by democratizing treatment and standardizing decision-making counseling, the decision aid can mediate attitudes and reduce stigma. The investigators hypothesize by delivering standardized, high-quality knowledge to both provider and patient, that stigma can be reduced in both parties. In Aim 1 the investigators will adapt an existing decision aid for OUD treatment to the specific context of rural hospital care. This decision aid will be a part of an existing bundled care program for OUD and related infections that the investigators have implemented in these hospitals. In Aim 2 the investigators will conduct a randomized pilot comparing the decision aid intervention with counseling as usual without decision aid to assess feasibility, acceptability and preliminary effectiveness for reducing stigma in substance use, HIV, OUD pharmacotherapy and harm reduction. The investigators will measure these around the time of the intervention and in longitudinal follow up. The findings could potentially identify a novel intervention and methodology for treatment expansion and stigma reduction that has not been previously explored, especially in the rural context, where need is high. Following the successful completion of this pilot trial, the investigators will develop an expanded multi-site comparative effectiveness trial of the decision aid, implementation studies, and cost-effectiveness analysis.

ELIGIBILITY:
Inclusion Criteria:

* Patients from a rural community currently admitted or recently admitted to Barnes-Jewish Hospital
* Admission must be for an infection associated with intravenous drug use
* Patient must be willing to speak with healthcare provider about medications for opioid use disorder (MOUDs)
* patient must be over 18 years old
* must be able to complete electronic survey written in English

Exclusion Criteria:

* None

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2022-04-07 (Actual); Primary Completion 2024-03-31 (Actual); Study Completion 2024-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael J. Durkin, MD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Barnes Jewish Hospital, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Baseline Counseling As Usual - Patient | Shared Decision Making Aid - Patient | Baseline Counseling As Usual - Provider | Shared Decision Making Aid - Provider
Started | 23 | 23 | 7 | 9
Completed | 23 | 23 | 7 | 9
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Baseline Counseling As Usual - Patient | Shared Decision Making Aid - Patient | Baseline Counseling As Usual - Provider | Shared Decision Making Aid - Provider | Total
Number analyzed (Participants) | 23 | 23 | 7 | 9 | 62
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 23 | 23 | 7 | 9 | 62
  >=65 years | 0 | 0 | 0 | 0 | 0
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 35 [31 to 44] | 35 [32 to 42] | 34 [29 to 41.5] | 38 [35 to 47] | 35 [31 to 43]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 14 | 7 | 6 | 40
  Male | 10 | 9 | 0 | 3 | 22
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 2 | 0 | 1 | 3
  White | 22 | 18 | 4 | 6 | 50
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 3 | 3 | 2 | 9
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 23 | 23 | 7 | 9 | 62

OUTCOME MEASURES:

1. Primary Outcome: Patient Internalized Stigma Towards Medicaid for Opioid Use Disorder (MOUDs) Over the Course of the Project
Description: Sum of 6 5-point Likert scale questions that determines self-reported stigma on taking MOUDs. This was compromised of 6 separate questions with a scale of 1-5 with 1 having the lowest stigma and 5 having the highest stigma. The range is thus 6 - 30.
Time Frame: 3 months
Population: Number of participants recruited and enrolled
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Baseline Counseling As Usual - Patient | Shared Decision Making Aid - Patient
Number analyzed (Participants) | 23 | 23
score on a scale
  Baseline | 15 [6 to 25] | 11 [6 to 27]
  Immediate follow-up | 14 [6 to 29] | 8 [6 to 24]
  2 week post-discharge | 8 [6 to 21] | 7 [6 to 23]
  90 days post-discharge | 8 [6 to 25] | 9 [6 to 17]
Statistical Analysis 1: Comparison: Baseline Counseling As Usual - Patient vs Shared Decision Making Aid - Patient; Test type: Other — Mann-Whitney U; p = 0.32, Wilcoxon (Mann-Whitney); Mann-Whitney U = 0.32
Statistical Analysis 2: Comparison: Baseline Counseling As Usual - Patient; Baseline survey compared with immediate follow-up survey; Test type: Other — Mann-Whitney U; p = 0.39, Wilcoxon (Mann-Whitney); Mann-Whitney U = 0.39
Statistical Analysis 3: Comparison: Baseline Counseling As Usual - Patient; 2 weeks post-discharge compared with baseline survey; Test type: Other — Mann-Whitney U; p = 0.21, Wilcoxon (Mann-Whitney); Mann-Whitney U = 0.21
Statistical Analysis 4: Comparison: Baseline Counseling As Usual - Patient; 90 days post-discharge compared with baseline survey; Test type: Other; p = 0.19, Wilcoxon (Mann-Whitney); Mann-Whitney U = 0.19
Statistical Analysis 5: Comparison: Shared Decision Making Aid - Patient; Baseline survey versus immediate follow-up; Test type: Other; p = 0.38, Wilcoxon (Mann-Whitney); Mann-Whitney U = 0.38
Statistical Analysis 6: Comparison: Shared Decision Making Aid - Patient; 2 weeks post-discharge compared with baseline survey; Test type: Other; p = 0.25, Wilcoxon (Mann-Whitney); Mann-Whitney U = 0.25
Statistical Analysis 7: Comparison: Shared Decision Making Aid - Patient; 90 days post-discharge compared with baseline survey; Test type: Other; p = 0.07, Wilcoxon (Mann-Whitney); Mann-Whitney U = 0.07
Statistical Analysis 8: Comparison: Baseline Counseling As Usual - Patient vs Shared Decision Making Aid - Patient; Immediate follow-up between the two arms; Test type: Other; p = 0.03, Wilcoxon (Mann-Whitney); Mann-Whitney U = 0.03
Statistical Analysis 9: Comparison: Baseline Counseling As Usual - Patient vs Shared Decision Making Aid - Patient; 2 weeks post-discharge comparison between the 2 arms; Test type: Other; p = 0.65, Wilcoxon (Mann-Whitney); Mann-Whitney U = 0.65
Statistical Analysis 10: Comparison: Baseline Counseling As Usual - Patient vs Shared Decision Making Aid - Patient; 90-days post discharge compared between the 2 arms; Test type: Other; p = 0.97, Wilcoxon (Mann-Whitney); Mann-Whitney U = 0.97

2. Secondary Outcome: Patient Anticipated MOUD Stigma
Description: This 5-point Likert scale was compromised of 7 questions of a range of 7-35. The lower score denotes the lower stigma and the higher score denotes the higher stigma.
Time Frame: 3 months
Population: The Mann-Whitney U test was used to analyze anticipated MOUD stigma.
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Baseline Counseling As Usual - Patient | Shared Decision Making Aid - Patient
Number analyzed (Participants) | 23 | 23
score on a scale
  Baseline | 20 [7 to 34] | 21 [7 to 32]
  Immediate follow-up | 19 [7 to 32] | 17 [7 to 35]
  2 weeks post-discharge | 18 [10 to 25] | 13 [7 to 29]
  90 days post-discharge | 11 [7 to 30] | 14 [7 to 30]
Statistical Analysis 1: Comparison: Baseline Counseling As Usual - Patient vs Shared Decision Making Aid - Patient; Baseline comparison between the 2 arms; Test type: Other; p = 0.77, Wilcoxon (Mann-Whitney); Mann-Whitney U = 0.77
Statistical Analysis 2: Comparison: Baseline Counseling As Usual - Patient; Immediate follow-up compared with baseline survey; Test type: Other; p = 0.85, Wilcoxon (Mann-Whitney); Mann-Whitney U = 0.85
Statistical Analysis 3: Comparison: Baseline Counseling As Usual - Patient; 2-week post-discharge compared with baseline survey; Test type: Other; p = 0.38, Wilcoxon (Mann-Whitney); Mann-Whitney U = 0.38
Statistical Analysis 4: Comparison: Baseline Counseling As Usual - Patient; 90-day post discharge compared with baseline survey; Test type: Other; p = 0.21, Wilcoxon (Mann-Whitney); Mann-Whitney U = 0.21
Statistical Analysis 5: Comparison: Shared Decision Making Aid - Patient; Immediate follow-up compared with baseline survey; Test type: Other; p = 0.32, Wilcoxon (Mann-Whitney); Mann-Whitney U = 0.32
Statistical Analysis 6: Comparison: Shared Decision Making Aid - Patient; 2 week post-discharge compared with baseline survey; Test type: Other; p = 0.09, Wilcoxon (Mann-Whitney); Mann-Whitney U = 0.09
Statistical Analysis 7: Comparison: Shared Decision Making Aid - Patient; 90-day post-discharge compared with baseline survey; Test type: Other; p = 0.07, Wilcoxon (Mann-Whitney); Mann-Whitney U = 0.07
Statistical Analysis 8: Comparison: Baseline Counseling As Usual - Patient vs Shared Decision Making Aid - Patient; 2 weeks post-discharge compared between the 2 arms; Test type: Other; p = 0.26, Wilcoxon (Mann-Whitney); Mann-Whitney U = 0.26
Statistical Analysis 9: Comparison: Baseline Counseling As Usual - Patient vs Shared Decision Making Aid - Patient; Immediate follow-up compared between the 2 arms; Test type: Other; p = 0.69, Wilcoxon (Mann-Whitney); Mann-Whitney U = 0.69
Statistical Analysis 10: Comparison: Baseline Counseling As Usual - Patient vs Shared Decision Making Aid - Patient; 90-day post-discharge compared between the 2 arms; Test type: Other; p = 0.32, Wilcoxon (Mann-Whitney); Mann-Whitney U = 0.32

3. Secondary Outcome: Patient Satisfaction With Clarity of Shared Decision Aid
Description: Likert scale from 1-4 with 1 being the best and 4 being the worst. There is no statistical analysis for this secondary outcome as patients who did not receive the decision aid cannot provide satisfaction regarding clarity of shared decision aid.
Time Frame: Immediate post-baseline survey
Population: Mann-Whitney U
Measure: Mean (Full Range); unit: score on a scale
Groups:
- Shared Decision Making Aid: Patients randomized to the decision aid arm will receive all of the above as well as a shared decision making aid. This will be a 10-minute tablet- or web-based intervention administered by one of our wraparound care service team members in-person or via telehealth (or possibly in person depending on pandemic procedures). IT will be a 10-minute procedure with summary of decision considerations and patient value assessment.The provider will have access to then have access to this summary in making final care decisions with the patient.
Arm/Group | Shared Decision Making Aid
Number analyzed (Participants) | 18
score on a scale | 1.33 [1 to 2]

4. Secondary Outcome: Patient Satisfaction With Helpfulness of Shared Decision Aid
Description: Likert scale from 1-4 with 1 being the best and 4 being the worst
Time Frame: Immediate post-baseline survey
Population: Mann-Whitney U
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Shared Decision Making Aid
Number analyzed (Participants) | 18
score on a scale | 1.44 [1 to 3]

5. Secondary Outcome: Overall Patient Satisfaction With the Shared Decision Aid
Description: "I like the decision aid", "The decision aid is appealing", "The decision aid is easy to use", and "The decision aid is doable". The scale range is 1 to 2 with a score of 1 being a better outcome.
Time Frame: Immediate post-baseline survey
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Shared Decision Making Aid
Number analyzed (Participants) | 18
score on a scale
  I like the decision aid | 1.06 [1 to 2]
  The decision aid is appealing | 1.06 [1 to 2]
  The decision aid is easy to use | 1.06 [1 to 2]
  The decision aid is doable | 1 [1 to 1]

6. Secondary Outcome: Provider Willingness To Work With Patients With Opioid Use Disorder
Description: 5-point Likert scale where score of 1 is the most stigma and 5 is the least stigma. The overall number is a sum of 4 questions with a theoretical range of 4 - 20.
Time Frame: Immediately post-intervention
Population: Healthcare providers taking care of patients with Opioid Use Disorder
Measure: Median (Full Range); unit: score on a scale
Groups:
- Assessing Stigma of Providers of Patients Randomized to Shared Decision Aid: Providers who provide care for patients enrolled in this project will be asked to participate in a survey to assess their stigma in regards to taking care of patients with opioid use disorder. This will be a 10-minute tablet- or web-based in-person survey administered by one of our wraparound care service team members. These healthcare providers were matched with a patient who was randomized to the shared decision aid for opioid use disorder.
- Assessing Stigma of Providers of Patients Randomized to Standard Care: Providers who provide care for patients enrolled in this project will be asked to participate in a survey to assess their stigma in regards to taking care of patients with opioid use disorder. This will be a 10-minute tablet- or web-based in-person survey administered by one of our wraparound care service team members. These healthcare providers were matched with a patient who was randomized to the standard clinical care for opioid use disorder.
Arm/Group | Assessing Stigma of Providers of Patients Randomized to Shared Decision Aid | Assessing Stigma of Providers of Patients Randomized to Standard Care
Number analyzed (Participants) | 9 | 7
score on a scale
  Baseline | 20 [5 to 20] | 20 [17 to 20]
  Immediate follow-up post randomization of patient | 20 [5 to 20] | 20 [20 to 20]
Statistical Analysis 1: Comparison: Assessing Stigma of Providers of Patients Randomized to Shared Decision Aid vs Assessing Stigma of Providers of Patients Randomized to Standard Care; Test type: Other — Mann-Whitney U; p = 1.00, Wilcoxon (Mann-Whitney); Mann-Whitney U = 1.00
Statistical Analysis 2: Comparison: Assessing Stigma of Providers of Patients Randomized to Shared Decision Aid; Test type: Other — Mann-Whitney U; p = 1.00, Wilcoxon (Mann-Whitney); Mann-Whitney U = 1.00
Statistical Analysis 3: Comparison: Assessing Stigma of Providers of Patients Randomized to Standard Care; Test type: Other — Mann-Whitney U; p = 0.12, Wilcoxon (Mann-Whitney); Mann-Whitney U = 0.12
Statistical Analysis 4: Comparison: Assessing Stigma of Providers of Patients Randomized to Shared Decision Aid vs Assessing Stigma of Providers of Patients Randomized to Standard Care; Immediate follow-up; Test type: Other — Mann-Whitney U; p = 0.12, Wilcoxon (Mann-Whitney); Mann-Whitney U = 0.12

7. Secondary Outcome: Hospital Policy Stigma Towards Patients With Opioid Use Disorder
Description: 5-point Likert scale where score of 1 least stigma towards patients with opioid use disorder and 5 is the highest stigma towards patients with opioid use disorder. The overall number is a sum of 4 questions with a theoretical range of 4 - 20.
Time Frame: Immediate
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Assessing Stigma of Providers of Patients Randomized to Shared Decision Aid | Assessing Stigma of Providers of Patients Randomized to Standard Care
Number analyzed (Participants) | 9 | 7
score on a scale
  Baseline | 8 [4 to 10] | 7 [5 to 9]
  Immediate follow-up post patient randomization | 7 [4 to 13] | 7 [4 to 8]
Statistical Analysis 1: Comparison: Assessing Stigma of Providers of Patients Randomized to Shared Decision Aid vs Assessing Stigma of Providers of Patients Randomized to Standard Care; Test type: Other — Mann-Whitney U; p = 0.48, Wilcoxon (Mann-Whitney); Mann-Whitney U = 0.48
Statistical Analysis 2: Comparison: Assessing Stigma of Providers of Patients Randomized to Shared Decision Aid; Test type: Other — Mann-Whitney U; p = 1.00, Wilcoxon (Mann-Whitney); Mann-Whitney U = 1.00
Statistical Analysis 3: Comparison: Assessing Stigma of Providers of Patients Randomized to Standard Care; Test type: Other — Mann-Whitney U; p = 0.17, Wilcoxon (Mann-Whitney); Mann-Whitney U = 0.17
Statistical Analysis 4: Comparison: Assessing Stigma of Providers of Patients Randomized to Shared Decision Aid vs Assessing Stigma of Providers of Patients Randomized to Standard Care; Immediate follow-up; Test type: Other — Mann-Whitney U; p = 0.42, Wilcoxon (Mann-Whitney); Mann-Whitney U = 0.42

8. Secondary Outcome: Provider Comfort Treating Patients With Opioid Use Disorder
Description: A 6 question 5-point Likert scale with a scale of 1= least stigma and 5=most stigma. A total of 6 questions were asked. Thus the range is 6 - 30.
Time Frame: Immediate post-intervention
Population: Healthcare providers who care of patients with opioid use disorder
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Assessing Stigma of Providers of Patients Randomized to Shared Decision Aid | Assessing Stigma of Providers of Patients Randomized to Standard Care
Number analyzed (Participants) | 9 | 7
score on a scale
  Baseline | 17 [15 to 20] | 17 [16 to 20]
  Immediate follow-up post patient randomization | 18 [15 to 30] | 18 [15 to 19]
Statistical Analysis 1: Comparison: Assessing Stigma of Providers of Patients Randomized to Shared Decision Aid vs Assessing Stigma of Providers of Patients Randomized to Standard Care; Baseline; Test type: Other — Mann-Whitney U; p = 1.00, Wilcoxon (Mann-Whitney); Mann-Whitney U = 1.00
Statistical Analysis 2: Comparison: Assessing Stigma of Providers of Patients Randomized to Shared Decision Aid; Baseline versus immediate follow-up; Test type: Other — Mann-Whitney U; p = 0.11, Wilcoxon (Mann-Whitney); Mann-Whitney U = 0.11
Statistical Analysis 3: Comparison: Assessing Stigma of Providers of Patients Randomized to Standard Care; Baseline versus immediate follow-up; Test type: Other — Mann-Whitney U; p = 0.89, Wilcoxon (Mann-Whitney); Mann-Whitney U = 0.89
Statistical Analysis 4: Comparison: Assessing Stigma of Providers of Patients Randomized to Shared Decision Aid vs Assessing Stigma of Providers of Patients Randomized to Standard Care; Immediate follow-up; Test type: Other — Mann-Whitney U; p = 0.55, Wilcoxon (Mann-Whitney); Mann-Whitney U = 0.55

9. Secondary Outcome: Provider Stigma Towards Patients With Opioid Use Order
Description: as for outcome 8
Time Frame: Immediate
Population: Healthcare providers who treat patients with opioid use disorder
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Assessing Stigma of Providers of Patients Randomized to Shared Decision Aid | Assessing Stigma of Providers of Patients Randomized to Standard Care
Number analyzed (Participants) | 9 | 7
score on a scale
  Baseline | 14 [11 to 16] | 14 [12 to 15]
  Immediate follow-up post patient randomization | 14 [12 to 19] | 13 [12 to 14]
Statistical Analysis 1: Comparison: Assessing Stigma of Providers of Patients Randomized to Shared Decision Aid vs Assessing Stigma of Providers of Patients Randomized to Standard Care; Baseline; Test type: Other — Mann-Whitney U; p = 0.66, Wilcoxon (Mann-Whitney); Mann-Whitney U = 0.66
Statistical Analysis 2: Comparison: Assessing Stigma of Providers of Patients Randomized to Shared Decision Aid; Baseline versus immediate follow-up post randomization; Test type: Other — Mann-Whitney U; p = 0.20, Wilcoxon (Mann-Whitney); Mann-Whitney U = 0.20
Statistical Analysis 3: Comparison: Assessing Stigma of Providers of Patients Randomized to Standard Care; Baseline versus immediate follow-up post randomization; Test type: Other — Mann-Whitney U; p = 0.85, Wilcoxon (Mann-Whitney); Mann-Whitney U = 0.85
Statistical Analysis 4: Comparison: Assessing Stigma of Providers of Patients Randomized to Shared Decision Aid vs Assessing Stigma of Providers of Patients Randomized to Standard Care; Immediate follow-up post randomization; Test type: Other — Mann-Whitney U; p = 0.07, Wilcoxon (Mann-Whitney); Mann-Whitney U = 0.07

ADVERSE EVENTS:
Time Frame: Participants were followed for 3 months for any adverse events.
Arm/Group | Baseline Counseling As Usual - Patient | Shared Decision Making Aid - Patient | Baseline Counseling As Usual - Provider | Shared Decision Making Aid - Provider
All-Cause Mortality (participants affected / at risk) | 1/23 | 1/23 | 0/7 | 0/9
Serious Adverse Events (participants affected / at risk) | 1/23 | 2/23 | 0/7 | 0/9
Other Adverse Events (participants affected / at risk) | 0/23 | 0/23 | 0/7 | 0/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Baseline Counseling As Usual - Patient (N=23) | Shared Decision Making Aid - Patient (N=23) | Baseline Counseling As Usual - Provider (N=7) | Shared Decision Making Aid - Provider (N=9)
Overdose (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) — Drug overdose unrelated to survey
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Pneumonia unrelated to survey

LIMITATIONS AND CAVEATS:
Our preliminary findings included patients who were hospitalized. Anecdotally ,our team needed time to screen, recruit, and consent participants. On average, this ended up taking about 2 days. Our findings were biased more towards individuals who were hospitalized for a prolonged period of time and for individuals with a long history of opioid use disorder. If or how this would work in outpatient settings needs to be evaluated. The shared decision aid was somewhat time consuming to complete.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol and Statistical Analysis Plan (2022-03-25): https://cdn.clinicaltrials.gov/large-docs/12/NCT05352412/Prot_SAP_000.pdf
  • Informed Consent Form: Patient Letter of Consent (2022-03-25): https://cdn.clinicaltrials.gov/large-docs/12/NCT05352412/ICF_001.pdf
  • Informed Consent Form: Provider Letter of Consent (2022-04-04): https://cdn.clinicaltrials.gov/large-docs/12/NCT05352412/ICF_002.pdf